CLINICAL TRIAL: NCT01007318
Title: Prospective, Randomized Study of Single Port and Conventional Laparoscopic Appendectomy in Acute Appendicitis
Brief Title: Safety and Efficacy Study of Single Port Laparoscopic Appendectomy in Acute Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: KyungHee University School of Medicine, Korea (Unknown)
Responsible Party: Principal Investigator, Byung Mo Kang, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: khnmc IRB 2009-026
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single port (Active Comparator): Single port through the transumbilical incision was made by wound retractor combined with surgical glove and then 3 trocal was inserted to the finger part of the surgical glove. Laparoscopic instrument was working through the single port and resected appendix removed through it.
  Interventions: Procedure: Single port laparoscopic appendectomy
- 3 port (Active Comparator): 3 port laparoscopic appendectomy was done by conventional method
  Interventions: Procedure: 3 port laparoscopic appendectomy

INTERVENTIONS:
Procedure: Single port laparoscopic appendectomy — Single port through the transumbilical 2-cm incision
  Other Names: single port laparoscopic surgery
  Arms: Single port
Procedure: 3 port laparoscopic appendectomy — 3 trocars was inserted in infraumbilical, left lower quadrant, and suprapubic area
  Other Names: conventional laparoscopic appendectomy
  Arms: 3 port

SUMMARY:
The aim of this study is to investigate the safety and efficacy of single port laparoscopic appendectomy compared with conventional laparoscopic appendectomy in adults with acute appendicitis.

DETAILED DESCRIPTION:
Laparoscopic appendectomy improved the postoperative functional outcomes in the treatment of acute appendectomy. In addition, recently single port laparoscopic surgery was introduced in the laparoscopy-dedicated center. When compared with conventional 3 port laparoscopic appendectomy, single port laparoscopic appendectomy was expected to be less painful, more rapid recovery of bowel function, and better cosmetic. In this prospective randomized trial, we tried to investigate the superiority of this new technique in adult patients with acute appendectomy.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed acute appendicitis

Exclusion Criteria:

* Age less than 7 or more than 75 years old
* Gangrenous appendicitis
* Combined generalized peritonitis
* ASA score more than 3 point
* Pregnant women
* Cases requiring draining tube

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety | 1 month
  30 day morbidity and mortality

SECONDARY OUTCOMES:
Efficacy | 1 day
  Operative time
Efficacy | 2 days
  Postoperative pain score
Efficacy | 2 days
  Postoperative functional recovery
Efficacy | 7 days
  Duration of postoperative hospital stay
Efficacy | 7 days
  Cost

CONTACTS AND LOCATIONS:
Overall Officials: Suk Hwan Lee, MD. PhD, Principal Investigator — Kyung Hee University School of Medicine
Locations (1):
- Kyung Hee University School of Medicine, Neo Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang BM, Choi SI, Kim BS, Lee SH. Single-port laparoscopic surgery in uncomplicated acute appendicitis: a randomized controlled trial. Surg Endosc. 2018 Jul;32(7):3131-3137. doi: 10.1007/s00464-018-6028-0. Epub 2018 Jan 16. PMID 29340826